CLINICAL TRIAL: NCT05017974
Title: Randomized Controlled Trial of Mindfulness-based Stress Reduction Plus Prenatal Sleep Supplement Versus Usual Care: Acceptability, Feasibility, and Adherence
Brief Title: Research on Improving Sleep During Pregnancy
Acronym: RISE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20-32853; K23AT009896 (NIH)
Record Dates: First submitted 2021-08-17; First posted 2021-08-24 (Actual); Results first posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Sleep; Pregnancy Related
Keywords: pregnancy; sleep; mindfulness
MeSH Terms: interventions — Mindfulness-Based Stress Reduction; Therapeutics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction plus Prenatal Sleep supplement (MBSR+PS) (Experimental): The study intervention is standard mindfulness-based stress reduction (MBSR), which will be delivered through 8 weekly 2.5-hour sessions via video conferencing to groups of 20-30 pregnant and non-pregnant people. MBSR also consists of a 2.5-hour orientation session, a 30-minute private interview with the instructor, and an all-day retreat, all conducted via video conferencing. The supplemental prenatal sleep content will be delivered through 6-8 30-minute sessions via video conferencing either individually or to small groups, and draws material from mindfulness-based therapy for insomnia, mindfulness-based childbirth and parenting program, and cognitive behavior therapy for prenatal insomnia.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction plus Prenatal Sleep supplement; Other: Treatment as Usual
- Treatment as Usual (Other): The control condition was designed to reflect standard care for insomnia patients. No limits are placed on receiving non-study treatment, including medication or psychotherapy, with the exception of asking participants to refrain from participating in non-study mindfulness practice. Use of non-study treatment will be tracked.
  Interventions: Other: Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction plus Prenatal Sleep supplement — MBSR+PS
  Arms: Mindfulness-Based Stress Reduction plus Prenatal Sleep supplement (MBSR+PS)
Other: Treatment as Usual — TAU

SUMMARY:
The overarching goal is to utilize a randomized control design to examine acceptability, feasibility, and adherence of mindfulness-based stress reduction plus prenatal sleep supplement (MBSR+PS) compared to treatment as usual among pregnant people with poor sleep quality (n=50).

DETAILED DESCRIPTION:
Poor sleep quality is highly prevalent during pregnancy, with important implications for maternal and infant health and well-being. Despite this, there is limited research on interventions to improve prenatal sleep, and prior research did not target the specific factors contributing to poor sleep quality in this population. Specifically, pregnant people report that physical symptoms, including discomfort and pain, disturb their sleep. In non-pregnant populations, this pain-sleep relationship is bidirectional, and maladaptive psychological responses to pain further exacerbate poor sleep. Theory and empirical evidence indicate that mindfulness-based interventions may be effective for targeting these psychological responses. The overarching goal is to utilize a randomized control design to examine acceptability, feasibility, and adherence of mindfulness-based stress reduction plus prenatal sleep supplement (MBSR+PS) compared to treatment as usual among pregnant people with poor sleep quality (n=50). Participants will be recruited to complete study questionnaires at two timepoints during pregnancy. Participants randomized to MBSR+PS will receive usual care, will be asked to attend 8 weekly group MBSR sessions (in addition to the MBSR orientation session, 1:1 interview with the instructor, and daylong retreat) and 6-8 PS sessions individually or in small groups, and will complete daily sleep and home practice diaries. Participants randomized to treatment as usual will receive usual care.

The specific aims are:

1. To determine acceptability of MBSR+PS.
2. To determine feasibility of MBSR+PS.
3. To determine adherence to MBSR+PS.
4. To explore evidence of change in psychological mediators.
5. To explore between-group differences in sleep.
6. To explore group differences in other critical clinical outcomes (e.g. depressive symptoms, anxiety symptoms, stress).

There is strong conceptual basis to predict the potential benefit of this approach for pregnant people. Targeting psychological responses to poor sleep during pregnancy may have significant public health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Pregnancy 12-28 weeks gestation at time of intervention start
* 18 years of age or older
* Regular access to a web-enabled computer, phone or tablet
* Ability to read and speak English, and to provide informed consent
* Poor sleep quality (PSQI > 5)

Exclusion Criteria:

* Self-reported sleep disorder (e.g. sleep apnea, narcolepsy, parasomnia, circadian rhythm disorder)
* Shift-work or nighttime caregiving responsibilities
* Psychological, medical, or other issues that necessitate priority treatment (e.g. active suicidality, probable depression (PHQ-9 ≥ 10), psychosis, on bed rest, multiple gestation)
* Current regular mindfulness practice (>20 minutes/week)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2021-09-08 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer N Felder, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Started | 26 | 26
Completed | 24 | 24
Not Completed | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual | Total
Number analyzed (Participants) | 26 | 26 | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.31 (5.02) | 31.85 (5.45) | 32.58 (5.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 26 | 52
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian, White, or European American | 13 | 16 | 29
  African American or Black | 4 | 3 | 7
  Latina, Latin American, or Hispanic | 3 | 2 | 5
  Asian or Pacific Islander | 6 | 3 | 9
  Bi- or multi-racial or -ethnic | 0 | 2 | 2
Pittsburgh Sleep Quality Index (PSQI) Score [Mean (Standard Deviation); unit: units on a scale] — The Pittsburgh Sleep Quality Index (PSQI) score ranges from 0 to 21. A total score of 5 or more indicates poor sleep quality; the higher the score, the worse the sleep quality.
  units on a scale | 7.12 (2.57) | 7.15 (1.74) | 7.13 (2.17)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Total Score Greater Than or Equal to 24 on the 8-item Client Satisfaction Questionnaire (CSQ-8) at 12 Weeks
Description: The Client Satisfaction Questionnaire (CSQ-8) score ranges from 8 to 32, with high scores indicating greater satisfaction. The CSQ-8 score of participants randomized to MBSR+PS will be reported; participants randomized to TAU will not complete the CSQ-8 as the questions pertain to the MBSR+PS program.
Time Frame: Post-intervention, an average of 12 weeks
Population: The overall number of participants analyzed (n=23) is one lower than reported in the participant flow module because one participant skipped the items for this measure but completed the majority of the other endpoint surveys.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS)
Number analyzed (Participants) | 23
Participants | 20

2. Secondary Outcome: Number of Participants Who Attend at Least One Session of MBSR and the PS Supplement From Baseline to 12 Weeks
Description: Participants can attend 0-8 sessions of MBSR and of PS.
Time Frame: Baseline to post-intervention, an average of 12 weeks
Population: This measure will only be collected for the MBSR+PS group; it is not applicable for participants randomized to TAU.
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS)
Number analyzed (Participants) | 26
Participants | 23

3. Secondary Outcome: Number of Participants Completing Endpoint Measures at 12 Weeks
Description: For a measure to be considered complete, at least 95% of items must be completed.
Time Frame: Post-intervention, an average of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
Participants | 24 | 24

4. Secondary Outcome: Completeness of Study Measures at Baseline and at 12 Weeks
Description: For a measure to be considered complete, at least 95% of items must be completed. Completeness of study measures at baseline and 12 weeks are combined (averaged); the percentage of measures completed across timepoints is reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Number; unit: percentage of measures completed
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
percentage of measures completed | 95.2 | 96.1

5. Secondary Outcome: Percentage of MBSR and PS Sessions Attended
Description: This measure will not be collected for participants randomized to TAU.
Time Frame: Baseline to post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of sessions attended
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS)
Number analyzed (Participants) | 26
percentage of sessions attended
  MBSR attendance | 80.00 (8.08)
  PS attendance | 82.00 (7.10)

6. Secondary Outcome: Frequency of Home Practices From Baseline to 12 Weeks
Description: Participants randomized to MBSR+PS will complete daily diaries reporting their formal and informal practices. Participants randomized to TAU will not complete this measure.
Time Frame: Baseline to post-intervention, an average of 12 weeks
Population: Participants randomized to MBSR+PS. The participant flow module lists n=24 analyzed because 24 participants completed endpoint measures. The overall number of participants analyzed for this measure is n=23 because the three participants who did not initiate MBSR+PS were not invited to complete this measure.
Measure: Mean (Standard Deviation); unit: percentage of days
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS)
Number analyzed (Participants) | 23
percentage of days
  MBSR Home Practice | 85.84 (17.99)
  PS Home Practice | 96.66 (4.19)

7. Secondary Outcome: Duration of Home Practices From Baseline to 12 Weeks
Description: Participants randomized to MBSR+PS will complete daily diaries reporting their formal and informal practices. Participants assigned to TAU will not complete this measure.
Time Frame: Baseline to post-intervention, an average of 12 weeks
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: number of minutes per day
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS)
Number analyzed (Participants) | 23
number of minutes per day | 36.21 (35.00)

8. Secondary Outcome: Change in Self Compassion Scale - Short Form (SCS-SF) From Baseline to 12 Weeks
Description: The Self Compassion Scale - Short Form (SCS-SF) score ranges from 1 to 5, with higher scores indicating greater self-compassion. The change in SCS-SF score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | 1.12 (5.64) | 2.71 (7.57)

9. Secondary Outcome: Change in Five-Facet Mindfulness Questionnaire (FFMQ) Nonjudging and Nonreactivity Factors From Baseline to 12 Weeks
Description: We included two factors of the Five-Facet Mindfulness Questionnaire (FFMQ): the nonjudging factor (score ranges from 8 to 40) and the non-reactivity factors (score ranges from 7 to 35). Higher scores indicate greater mindfulness. The change in factor scores from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale
  Nonjudging score | 2.00 (4.17) | 1.58 (5.72)
  Nonreacting score | 2.04 (5.15) | 1.46 (4.20)

10. Secondary Outcome: Change in Coping Strategies Questionnaire - Revised (CSQ-R) From Baseline to 12 Weeks
Description: The Coping Strategies Questionnaire - Revised (CSQ-R) score ranges from 0 to 36 on each of the 7 subscales, with higher scores indicating greater use of a coping strategy. The change in CSQ score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale
  Distracting score | .38 (.73) | -.09 (.98)
  Catastrophizing score | -.36 (.58) | -.14 (1.04)
  Ignoring score | -.25 (1.03) | .03 (1.21)
  Distancing score | .54 (1.34) | .41 (.98)
  Coping score | -.08 (.93) | -.05 (.97)
  Praying score | .04 (.95) | .33 (1.09)

11. Secondary Outcome: Change in Rumination-Reflection Questionnaire (RRQ) From Baseline to 12 Weeks
Description: The Rumination-Reflection Questionnaire (RRQ) score ranges from 12 to 60 for each of the two factors. Greater scores indicate greater tendency to ruminate and reflect. The change in RRQ score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale
  Rumination score | -1.46 (6.85) | -2.75 (5.84)
  Reflection score | .96 (3.85) | -.13 (5.04)

12. Secondary Outcome: Change in Pittsburgh Sleep Quality Index Score (PSQI) From Baseline to 12 Weeks
Description: The Pittsburgh Sleep Quality Index (PSQI) score ranges from 0 to 21. A total score of 5 or more indicates poor sleep quality; the higher the score, the worse the sleep quality. The change in PSQI score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | -2.58 (2.21) | -1.79 (2.06)

13. Secondary Outcome: Change in Insomnia Severity Index Score (ISI) From Baseline to 12 Weeks
Description: The Insomnia Severity Index (ISI) score ranges from 0 to 28, with higher scores indicating greater insomnia severity. The change in ISI score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | -5.29 (4.09) | -4.17 (4.06)

14. Secondary Outcome: Change in Dysfunctional Beliefs About Sleep Score (DBAS) From Baseline to 12 Weeks
Description: The Dysfunctional Beliefs About Sleep (DBAS) score ranges from 0 to 10, with a score of 4 or greater indicating unrealistic expectations for sleep, and greater scores indicating more dysfunctional beliefs about sleep. The change in DBAS score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | -1.11 (1.15) | -.96 (1.24)

15. Secondary Outcome: Change in Measures for Coping With Sleep Disturbances Score From Baseline to 12 Weeks
Description: The Measures for coping with sleep disturbances score ranges from 0 to 11, with greater scores indicating greater use of active coping measures for sleep disturbance. The change in Measures for coping with sleep disturbances score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Population: Data were not collected for this measure.
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 0 | 0

16. Secondary Outcome: Worry About Sleep Duration
Description: Single item measure that assesses whether participants worried about not getting enough sleep in the past 2 weeks.
Time Frame: Post-intervention, an average of 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 24 | 24
Participants | 9 | 8

17. Secondary Outcome: Change in Patient Health Questionnaire-9 Score (PHQ-9) From Baseline to 12 Weeks
Description: The Patient Health Questionnaire-9 (PHQ-9) score ranges from 0 to 27, with a score greater than or equal to 10 indicating moderate to severe depression, and the higher the score, the greater the depressive symptom severity. The change in PHQ-9 score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline to post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | -1.78 (2.70) | -1.38 (3.02)

18. Secondary Outcome: Change in PROMIS 6-item Anxiety Score From Baseline to 12 Weeks
Description: The PROMIS 6-item anxiety score ranges from 6 to 30, with higher scores indicating more severe anxiety; from raw scores, standardized T-scores can be determined. The change in PROMIS 6-item anxiety T-score from baseline to post-intervention (at 12 weeks) will be reported. The T-score values have a mean = 50 and SD = 10, with higher scores indicating greater anxiety.
  The T-scores are interpreted as follows:
  Less than 55 = None to slight anxiety 55.0-59.9 = Mild anxiety 60.0-69.9 = Moderate anxiety 70 and over = Severe anxiety
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
T-score | -1.45 (7.79) | -2.32 (7.55)

19. Secondary Outcome: Change in Perceived Stress Scale Score (PSS) From Baseline to 12 Weeks
Description: The Perceived Stress Scale score ranges from 0 to 40, with higher scores indicating greater appraisal of stress. The change in PSS score from baseline to post-intervention (at 12 weeks) will be reported.
Time Frame: Baseline and post-intervention, an average of 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
Number analyzed (Participants) | 26 | 26
units on a scale | -1.83 (3.93) | -2.46 (5.14)

ADVERSE EVENTS:
Time Frame: Baseline to 12 weeks
Arm/Group | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 8/26 | 7/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mindfulness-Based Stress Reduction Plus Prenatal Sleep Supplement (MBSR+PS) (N=26) | Treatment as Usual (N=26)
gestational diabetes dx (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
COVID diagnosis (Infections and infestations) | 3 (3) | 2 (2)
Elevated anxiety symptoms (Psychiatric disorders) | 2 (2) | 0 (0)
Elevated depressive symptoms (Psychiatric disorders) | 1 (1) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
High blood pressure (Cardiac disorders) | 1 (1) | 0 (0)
Passive suicidal ideation (Psychiatric disorders) | 1 (1) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT05017974/Prot_SAP_002.pdf